CLINICAL TRIAL: NCT00133731
Title: A Multinational, Randomized, Double-Blind, Double-Dummy, Exploratory, Parallel Group, Dose-Ranging Phase II Study to Evaluate Pharmacodynamics, Safety and Tolerability, and Pharmacokinetics of Several Intravenous Regimens of Factor Xa Inhibitor Otamixaban (XRP0673), in Comparison to Intravenous Unfractionated Heparin, in Subjects Undergoing Non-Urgent Percutaneous Coronary Intervention
Brief Title: The SEPIA-PCI Trial: Otamixaban in Comparison to Heparin in Subjects Undergoing Non-Urgent Percutaneous Coronary Intervention
Acronym: SEPIA-PCI
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: ICD Study Director, sanofi-aventis
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DRI6199; XRP0673
Record Dates: First submitted 2005-08-23; First posted 2005-08-24 (Estimated); Last update posted 2008-07-02 (Estimated); Status verified 2008-06

CONDITIONS: Angioplasty, Transluminal, Percutaneous Coronary
MeSH Terms: interventions — otamixaban; Heparin; Percutaneous Coronary Intervention

INTERVENTIONS:
Drug: Otamixaban (XRP0673)
Drug: Unfractionated Heparin
Procedure: Percutaneous Coronary Intervention

SUMMARY:
The objective of this dose-ranging study is to determine the effects of several intravenous (IV) regimens of otamixaban on pharmacodynamic markers (including markers of thrombosis and coagulation markers), safety/tolerability, clinical efficacy and pharmacokinetics.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Due to undergo non-urgent percutaneous coronary intervention (PCI)
* Planned treatment with aspirin and clopidogrel

Exclusion Criteria:

* Recent acute coronary syndrome
* Patients at risk for, or with prior recent, bleeding
* Patients have received recent prior treatment with an anticoagulant
* Creatinine clearance > 30 ml/min

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 947 (Actual)
Dates: Start 2004-09; Study Completion 2005-10 (Actual)

PRIMARY OUTCOMES:
Death, myocardial infarction, and urgent and non-urgent target vessel revascularization

SECONDARY OUTCOMES:
Bleeding events

CONTACTS AND LOCATIONS:
Overall Officials: ICD CSD, Study Director — Sanofi
Locations (89):
- United States (37):
  - Los Angeles Cardiology Associates, Los Angeles, California
  - Anil V. Shah, MD, Santa Ana, California
  - George Washington University Medical Faculty Associates, Washington D.C., District of Columbia
  - Florida Cardiovascular Research, Atlantis, Florida
  - Ocala Research Institute, Inc, Ocala, Florida
  - Central Florida Cardiology Group, PA, Orlando, Florida
  - Cardiology Associates, PA, Panama City, Florida
  - Heart Specialists of Sarasota, Sarasota, Florida
  - Cardiac Disease Specialists, Atlanta, Georgia
  - Emory University Hospital, Atlanta, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - Midwest Heart Foundation, Lombard, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Heart Care Midwest, Peoria, Illinois
  - Prairie Cardiovascular Consultants, Ltd, Springfield, Illinois
  - The Care Group, LLC, Indianapolis, Indiana
  - Iowa Heart Center, PC, Des Moines, Iowa
  - Kansas Cardiology Associates, Wichita, Kansas
  - UMass Memorial Medical Center, Worcester, Massachusetts
  - Minneapolis Heart Institute Foundation, Minneapolis, Minnesota
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - LeBauer Cardiovascular Research Foundation, Greensboro, North Carolina
  - Wake Heart Associates, Raleigh, North Carolina
  - The Lindner Clinical Trial Center, Cincinnati, Ohio
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - University of Oklahoma Health Science Center, Oklahoma City, Oklahoma
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Plaza Medical Group, PC, Oklahoma City, Oklahoma
  - Geisinger Clinic, Danville, Pennsylvania
  - Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - University of Pennsylvania Health System, Philadelphia, Pennsylvania
  - Columbia Heart Clinic, Columbia, South Carolina
  - Amarillo Heart Clinical Research Institute Inc, Amarillo, Texas
  - MEDVAMC, Houston, Texas
  - Audie Murphy VA Medical Center, San Antonio, Texas
  - Virginia Commonwealth University, Richmond, Virginia
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Belgium (2):
  - Cliniques Universitaires Saint-Luc, Brussels
  - UZ Gasthuisberg, Leuven
- Canada (9):
  - Foothills Medical Center, Calgary, Alberta
  - St. Boniface General Hospital, Winnipeg, Manitoba
  - Southlake Regional Health Centre, Newmarket, Ontario
  - Sunnybrook and Women's College Health Sciences Centre, Toronto, Ontario
  - Institut de Cardiologie de Montreal, Montreal, Quebec
  - Cardiac Catheterization Laboratories of the CHUM, Montreal, Quebec
  - CHUM - Hopital St-Luc, Montreal, Quebec
  - Hopital du Sacre-Coeur de Montreal, Montreal, Quebec
  - Centre Hospitalier Universitaire de Sherbrooke, Sherbrooke, Quebec
- Czechia (4):
  - University Hospital St Anna, Brno
  - University Hospital Hradec Kralove, Hradec Králové
  - General University Hospital, Prague
  - University Hospital Motol, Prague
- France (5):
  - Hopital Cardiologique Louis Pradel, Bron, Cedex
  - Institut Hospitalier Jacques Cartier, Massy, Cedex
  - Center Hospitalier Universitaire Jean-Minjoz, Besançon
  - Clinique Les Franciscaines, Nîmes
  - Institut de Cardiologie, Paris
- Germany (17):
  - Medisch Centrum Alkmarr, Alkmaar
  - Kerckhoff-Klinik GmbH, Bad Nauheim
  - Universitatmedizin Berlin, Berlin
  - Vivantes Klinikum Neukolln, Berlin
  - Virchow-Klinikum, Universtatsmedizin Berlin, Berlin
  - Klinikum der Universitat au Koln, Cologne
  - Krankanhaus Duren gem.GmbH, Düren
  - Klinikum der Johann Wolfgang Goethe-Universitat, Frankfurt
  - Universitatsklinikum Freiburg, Freiburg im Breisgau
  - Gamelinschalftspraxis, Hamburg
  - Universitatsklinikum Hamburg - Eppendorf, Hamburg
  - Klinikum der Friedrich-Schiller-Universitat Jena, Jena
  - Universitatsklinikum Schleswig-Holstein, Lübeck
  - Johannes Gutenberg Universitat Mainz, Mainz
  - Klinik der Universitat Munchen-Grobhadern, München
  - Klinikum Schwalmstadt der Schwalm-Eder-Kliniken, Schwalmstadt
  - Segeberger Kliniken GmbH, Segeberg
- Netherlands (5):
  - Amphia Hospital, Breda
  - Catherine Hospital, Eindhoven
  - St Antonius Hospital, Nieuwegein
  - Medisch Centrum Rijnmond-Zuid, Rotterdam
  - Isala Klinleken, Hospital De Weezenlanden, Zwolle
- Slovakia (2):
  - Middle Slovak Institute of Cardiovascular Diseases, Banská Bystrica
  - Slovak Institute of Cardiovascular Diseases, Bratislava
- South Africa (2):
  - Milpark Hospital, Johannesburg
  - Kuils River Private Hospital, Kuils River
- Spain (6):
  - Hospital San Juan de Alicante, Alicante
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital Universitari Bellvitge, Barcelona
  - Hospital Clinico San Carlos, Madrid
  - Hospital Gregorio Maranon, Madrid
  - Hospital Virgen de la Victoria, Málaga

REFERENCES:
- See also: Related Info — http://www.sanofi-aventis.com